CLINICAL TRIAL: NCT06365112
Title: The Endoscopic Surgical Technique of the Acetabulum: A Minimally Invasive Operative Technique for the Extraperitoneal Fixation of Acetabulum Fractures
Brief Title: Endoscopic Acetabulum Surgery
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21154
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Acetabulum Fracture
Keywords: acetabulum fracture; Endoscopy; Minimal invasive; collaboration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic assisted acetabulum fractrure treatment (Active Comparator)
  Interventions: Procedure: Endoscopy assisted
- Open reduction (Active Comparator)
  Interventions: Procedure: Endoscopy assisted

INTERVENTIONS:
Procedure: Endoscopy assisted — Endoscopy

SUMMARY:
Try to develop an endoscopic surgical technique to treat acetabulum fractures

DETAILED DESCRIPTION:
Endoscopically assisted acetabular fracture treatment

Introduction Acetabular fractures are uncommon trauma in Finnish population (1). The trauma mechanism usually in elderly population is fall in same level and in younger population high energy trauma such as motor vehicle accidents and fall from hights (1). Acetabular fractures are classified according the Letournel classification in which the fractures are divided in three main gategories: posterior column, both columns and anterior column (2).

These fractures are further divided into posterior column, posterior wall and posterior wall plus posterior column fractures. These posterior only fractures are usually operated through posterior approach. Both column fractures are further divided into six different types: transverse, transverse plus posterior wall, both column, T-shaped (posterior column and anterior hemitransverse), anterior column plus posterior hemitransverse; anterior wall plus posterior hemitransverse. Anterior approach is used usually to these fractures sometimes combined with posterior approach. The third fracture type is likewise divided into anterior column, anterior wall and anterior wall plus anterior column fractures, which are usually operated using anterior approach. (2)

Operative treatment is the golden standard in displaced high energy acetabulum fractures and technique has traditionally been open reduction and internal fixation (ORIF). Approach, which has been used to operate the anterior part of the acetabulum fractures, has been modified Stoppa in which the acetabulum is exposed through low midline incision in extraperitoneal region (3).

The problem with this approach is the visualization of the highest proportion of the pelvic brim and usually fractures highest point, because of the anatomical reasons, peritoneum and the arteria and vena femoralis goes nearby and sometimes prevent making the approach, reduction and plating of the fracture safely. Some patients have also post operative problems with the incision, they have pain in the anterior part of the pelvis. Also the dissection and sometimes detachment of the rectus abdominis muscles may cause serious problems post operatively.

Because of the problems with the approach, we have developed a novel technique in which we make the visibility with endoscopic technique. Extraperitoneal endoscopy is used commonly in the hernia reparation surgery nowadays (TEP). The acetabular fracture surgery is done in the same area as the hernia surgery so the approach itself is not a new method but the idea that fracture can be treated solely through endoroscopy is.

There are few published case reports similar as our method. One of which is from China and the technique was that they made endoscopic approacs and treated the fracture with 3D-printed model of the patients pelvis and then bended the plate matching the patients pelvis (4). The report is quite scarse and it lacks long term results altogether.

The other case report is from Germany and is otherwise similar as our technique, but they used additional ilioinguinal lateral approach to reduce the fracture and to introduce the plate. They state, that this method will be a standard procedure in future trauma management (5).

The reason for this study is thus to develop a novel method to operate anterior acetabular fractures endoscopically in cadavers and to test it in prospective matter in patients.

Aims of the study

* Develop a safe endoscopic surgical method to treat anterior acetabular fractures
* Test the method in patients prospectively
* To find out, if this novel method saves operation theatre time, blood loss, post operative patient satisfaction and VAS

Materials and methods The first part of the study includes the endoscopically assisted acetabular operation development in Tampere surgical education centre. The surgical method will be published.

The second part of the study is done in the Tampere University Hospital orthopaedics and traumatology ward. It consists of three (3) patients operated with this new method. In this part of the study, the patients will not be randomized, but we include all consecutive eligible patients. There will be at least one publication about this study part.

The third part of the study is done in randomized controlled study design in which the other group will be operated with the new endoscopically assisted method and the other group with the nowadays standard modified Stoppa approach. This study consist of ten (10) patients. There will be at least one publication about this study part.

Inclusion criteria are: age over 18 and anterior acetabular fracture, which can be treated with endoscopic method. Exclusion criteria are: age lower than 18 and previous lower abdomen operation

ELIGIBILITY:
Inclusion Criteria:

* Acetabulum fracture

Exclusion Criteria:

* <18years
* Previous lower abdominal operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with major complications | At three months
Number of patients with minor complications | At three months
Operation time | Intraoperative
Patient satisfaction using EQ5D | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided